CLINICAL TRIAL: NCT04830839
Title: Online Modules to Help Children Manage Medical Stress After an Injury: Recovery After Stress Toolkit (ReSeT) Pilot Study
Brief Title: Recovery After Stress Toolkit (ReSeT): Pilot Study
Acronym: ReSeT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Utah (Other); The University of Texas Health Science Center, Houston (Other); Tulane University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R24HD096350 (NIH)
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-12

CONDITIONS: Post-traumatic Stress Disorder
Keywords: post-traumatic stress; medical stress; e-health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This is a single group design as all eligible participants will be offered the 8 session Recovery after Stress Toolkit (ReSeT) program, including 8 self-guided child modules and 4 parent modules, as well as 8 parallel videoconferencing sessions with a therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recovery after Stress Toolkit (ReSeT) (Experimental): ReSeT is comprised of interactive web-based psychoeducational modules that are developmentally tailored for school age children (8-17 years) for use with synchronous e-health therapy sessions with a trained therapist.
  Participants in the ReSeT treatment will complete 8 modules and therapy sessions. Parents will also have access to 4 modules During the study, children/youth will be asked to complete all eight sessions of the online treatment together with the therapist over an 8 -12 week time period (to allow for scheduling/cancellations). For younger children, parents will participate in the beginning and end of each session. Sessions will last approximately 30-60 minutes and will occur approximately every week for an anticipated 4-8 hour time commitment. Parents of older children will be permitted to review the content independently and participate in feedback sessions.
  Interventions: Behavioral: Recovery after Stress Toolkit (ReSeT)

INTERVENTIONS:
Behavioral: Recovery after Stress Toolkit (ReSeT) — ReSeT involves online modules with parallel videoconferencing sessions. ReSeT integrates two evidence-based treatment methods: cognitive behavioral therapy coping skills (coping CBT) and direct exposure to trauma reminders through a trauma narrative.

SUMMARY:
Experiencing an accident and staying in the hospital can be scary and traumatic for children. The goal of this project is to develop an online resource to help children and their parents develop effective coping skills to manage their stress. Children ages 8-17 who exhibit signs of posttraumatic stress will view 8 online modules and attend weekly videoconferencing sessions with a therapist. Parents will have 4 modules to assist them in supporting their child after the injury.

DETAILED DESCRIPTION:
The overarching goal of this project is to provide a research and treatment resource for the management of psychological distress in children who have been hospitalized for a physical trauma. The investigators will pilot an innovative, brief e-health approach to treatment of PTSS designed to be delivered through the trauma system. The investigators will create interactive web-based psychoeducational modules that are developmentally tailored for school age children (8 to 17 years) for use with synchronous e-health therapy sessions with a trained therapist. Companion modules for parents will help parents to understand and respond to their child's PTSS. The investigators will perform a single-arm pilot trial of a brief e-health approach to treatment of PTSS (i.e., Recovery after Stress Toolkit; ReSeT). ( delete with usual care.)

ELIGIBILITY:
Inclusion Criteria:

* Ages of 8 to 17 years at time of enrollment
* Hospitalized for trauma at one of the following sites: PICU, ward or rapid treatment/observation unit (less than 23 hours stay)
* Both the parent and the child participating have the ability to read and speak English
* Have broadband internet availability at their home address
* Elevated post-traumatic stress symptoms (If the child exhibits clinically significant PTSS determined with the CPSS [Foa et al., 2001] with a score greater than or equal to 11 on the sum of the highest item by item score of parent/child report, they will be invited to participate in the pilot intervention. This methodology for using a joint score on the CPSS was informed by previous work indicating that both parents and children tend to underreport PTSS symptoms. Thus, implementing a multi-informant approach yields a more valid estimation of a child's psychopathology.)

Exclusion Criteria:

* Has sustained a moderate or severe TBI, as defined by a Glasgow Coma Score of less than 13
* Has been diagnosed with moderate or severe intellectual disability , low functioning autism spectrum disorder, or a developmental disability (This will be determined by medical chart review and confirmed with parent report: Has the child ever been diagnosed with an intellectual or developmental disability? i.e., child must be able to talk; the rationale for this is that they may have difficulty mastering the course content)
* Has a pre-existing severe psychiatric disorder that required prior psychiatric hospitalization (e.g., bipolar disorder, schizophrenia)
* The mechanism of the injury was abuse or interpersonal violence
* They are currently receiving psychotherapy
* Has been hospitalized for their injury for over 30 days
* No attempt will be made to recruit caregivers while their child is unstable, e.g. vitals are abnormal, there are major complications, or death may be imminent. Children with multiple injuries are eligible to participate but their caregivers will not be approached until any interventions (surgery, casting, etc.) are completed.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
The pilot is only anticipated to have 12-16 participants and thus,data may be identifiable. The investigators have decided to withhold the sharing individual participant data.

REFERENCES:
- [Background] Foa EB, Johnson KM, Feeny NC, Treadwell KR. The child PTSD Symptom Scale: a preliminary examination of its psychometric properties. J Clin Child Psychol. 2001 Sep;30(3):376-84. doi: 10.1207/S15374424JCCP3003_9. PMID 11501254
- [Background] Birmaher B, Brent DA, Chiappetta L, Bridge J, Monga S, Baugher M. Psychometric properties of the Screen for Child Anxiety Related Emotional Disorders (SCARED): a replication study. J Am Acad Child Adolesc Psychiatry. 1999 Oct;38(10):1230-6. doi: 10.1097/00004583-199910000-00011. PMID 10517055
- [Background] Varni JW, Magnus B, Stucky BD, Liu Y, Quinn H, Thissen D, Gross HE, Huang IC, DeWalt DA. Psychometric properties of the PROMIS (R) pediatric scales: precision, stability, and comparison of different scoring and administration options. Qual Life Res. 2014 May;23(4):1233-43. doi: 10.1007/s11136-013-0544-0. Epub 2013 Oct 2. PMID 24085345
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a tertiary care children's hospital with a Level I trauma center between late 2020 and early 2021.
Groups:
- Recovery After Stress Toolkit (ReSeT): ReSeT is comprised of interactive web-based psychoeducational modules that are developmentally tailored for school age children (8-17 years) for use with synchronous e-health therapy sessions with a trained therapist.
  Participants in the ReSeT treatment will complete 8 modules and therapy sessions. Parents will also have access to 4 modules During the study, children/youth will be asked to complete all eight sessions of the online treatment together with the therapist over an 8 -12 week time period (to allow for scheduling/cancellations). For younger children, parents will participate in the beginning and end of each session. Sessions will last approximately 30-60 minutes and will occur approximately every week for an anticipated 4-8 hour time commitment. Parents of older children will be permitted to review the content independently and participate in feedback sessions.
  Recovery after Stress Toolkit (ReSeT): ReSeT involves online modules with parallel videoconferencing sessions. ReSeT integrates two evidence-based treatment methods: cognitive behavioral therapy coping skills (coping CBT) and direct exposure to trauma reminders through a trauma narrative.
Period: Overall Study
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Adherence to the ReSeT intervention will be assessed by calculating the number of sessions participants complete out of the 8 proposed sessions.
Time Frame: Feasibility will be assessed at 12 weeks post-enrollment.
Measure: Mean (Full Range); unit: number of sessions completed
Units Other Than Participants: online sessions
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
Number analyzed (online sessions) | 48
number of sessions completed | 7.3 [6 to 8]

2. Primary Outcome: Acceptability
Description: The acceptability of the ReSeT intervention will be assessed with child and parent satisfaction surveys, and a qualitative interview with open-ended feedback about the program. The satisfaction surveys ask participants to rate their satisfaction with the program on a 4-point Likert scale (from "strongly disagree" to "strongly agree"), with higher scores indicative of greater satisfaction and acceptability. The ratio of child satisfactory responses over the total number of possible child satisfaction survey responses was calculated to measure overall child satisfaction.
Time Frame: Acceptability will be assessed at 12 weeks post-enrollment.
Measure: Number; unit: Satisfactory Survey Responses
Units Other Than Participants: Survey Responses
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
Number analyzed (Survey Responses) | 54
Satisfactory Survey Responses | 50

3. Primary Outcome: Length of Time to Complete Sessions
Description: The feasibility of the ReSeT intervention will be assessed with the number of weeks that it takes participants to complete the 8 sessions of the intervention. The intervention was designed to take place over a 12 week period, with sessions occurring weekly.
Time Frame: This outcome will be assessed at the end of the 8 sessions of the intervention.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 5
days | 65.2 (21.6)

4. Secondary Outcome: Child Post-traumatic Stress Symptoms (PTSS)
Description: The Child Post-Traumatic Stress Disorder Scale (CPSS; Foa et al, 2001) is a validated child report and parent proxy measure of PTSS. The measure is comprised of 24-items. The CPSS includes 17 questions mapping on to DSM-IV symptoms of PTSD rated on a 5-point scale that indicates how frequently each symptom occurs (0 = not at all, 1 = once a week or less/once in a while, 2 = 2 to 3 times a week/half the time, 3 = 4 to 5 times a week, 4=6 or more time a week/almost always). The minimum score for PTSS symptoms is 0 and the maximum is 80. A higher score indicates greater PTSS. The change in raw score from the 17 questions mapping PTSD symptoms was calculated from change in scores at 1 week post discharge to scores at 12 weeks post randomization.
Time Frame: Child PTSS from pre-intervention (within 6 months of the injury discharge) will be compared to the child's PTSS post-intervention, at 12 weeks post-enrollment or until the child has finished treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
score on a scale | -10 (10)

5. Secondary Outcome: Child Anxiety Symptoms
Description: The Screen Child Anxiety and Related Emotional Disorders (SCARED; Birmaher et al., 1999) is a widely used questionnaire that screens for anxiety and emotional disorders in children. The child self-report version will be used in this study, which consists of 41 items rated on a 3-point Likert scale ( 0 = not true or hardly ever true, 1 = somewhat true or sometimes true, 2 = very true or often true). This measures yields raw scores for anxiety disorder, panic disorder, generalized anxiety disorder, separation anxiety, social anxiety disorder, and significant school avoidance. Total scores range from 0-82, with scores above 25 indicating the presence of clinically significant anxiety. The change in total score from 1 week post discharge to 12 weeks post randomization was then calculated to get the overall change in score.
Time Frame: Child anxiety from pre-intervention (within 6 months of the injury discharge) will be compared to child anxiety post-intervention, at 12 weeks post-enrollment or until the child has finished treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
score on a scale | -7 (5)

6. Secondary Outcome: Child Quality of Life
Description: The Pediatric Quality of Life Inventory (PedsQL 4.0; Varni et al., 2001) is a well-validated parent- report measure consisting of 15 items that takes less than 5 minutes to complete. The PedsQL evaluates health-related quality of life by assessing the dimensions of physical, emotional, social, and cognitive functioning in children from infancy to 18 years of life age. The total quality of life scale score will be utilized. Scores range from 0-100, with higher scores indicating better health related quality of life. The Total quality of life score change from 1 week post discharge to 12 weeks post randomization was then calculated, with a greater change in total score indicating greater improvements in quality of life.
Time Frame: Child quality of life from pre-intervention (within 6 months of the injury discharge) will be compared to child quality of life post-intervention, at 12 weeks post-enrollment or until the child has finished treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
score on a scale | 9 (20)

7. Secondary Outcome: Child Depressive Symptoms
Description: The Patient Reported Outcomes Measurement Information System is a National Institutes of Health (NIH) initiative created to advance assessment of patient-reported outcomes. To measure child depressive symptoms for this outcome measure, the depression subscale t score (Mean 50 with SD 10) from the child reports were pulled, and the change in t score from 1 week post discharge to 12 weeks post randomization was calculated. As this outcome measure represents a change in t score from one time point to another, there is no standard minimum and maximum value to report. A greater change in t score represents a greater decrease in depressive symptoms, which represents better outcomes. There are no clinical cut-offs, however, greater than two standard deviations above or below the mean would represent an extreme value.
Time Frame: Child depressive symptoms from pre-intervention (within 6 months of the injury discharge) will be compared to child depressive symptoms post-intervention, at 12 weeks post-enrollment or until the child has finished treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Recovery After Stress Toolkit (ReSeT)
Number analyzed (Participants) | 6
score on a scale | -6 (7)

ADVERSE EVENTS:
Time Frame: from 1 week post discharge (start of study) to 12 weeks post randomization (or after completing 8 sessions for study)
Description: There were no adverse events reported.
Arm/Group | Recovery After Stress Toolkit (ReSeT)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT04830839/Prot_SAP_000.pdf